CLINICAL TRIAL: NCT01617148
Title: A Single Arm, Investigator Initiated Study of the Efficacy, Safety, and Tolerability of Intravitreal Aflibercept Injection in Subjects With Exudative Age-related Macular Degeneration Previously Treated With Ranibizumab or Bevacizumab (ASSESS Study)
Brief Title: Wet Macular Degeneration Study to Compare Ranibizumab or Bevacizumab to Aflibercept
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rishi Singh (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Rishi Singh, MD, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-AMD-1211
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Exudative Macular Degeneration
Keywords: Exudative Macular Degeneration; Aflibercept
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Aflibercept (Experimental): Subjects were given 2 mg (0.05 mL) of intravitreal aflibercept injection administered every month for the first 3 months, followed by 2 mg (0.05 mL) once every 2 months as per the drug label for the next 9 months.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Patients received 2 mg (0.05 mL) of intravitreal aflibercept injection administered monthly for the first 3 months, followed by 2 mg (0.05 mL) once every 2 months as per the drug label for the next 9 months.

SUMMARY:
This study will examine the use of Aflibercept in patients with exudative macular degeneration requiring intravitreal injections. Patients will be followed for 24 months. The follow up phase will be completed at month 36.

DETAILED DESCRIPTION:
The purpose of this study is to examine the use of Aflibercept in patients who have been previously treated with Ranibizumab or Bevacizumab for exudative macular degeneration. Specifically, we will examine its effect on macular degeneration, measured by SDOCT (Spectral Domain Optical Coherence Tomography) and ETDRS (Early Treatment Diabetic Retinopathy Study) visual acuity. This will be a prospective study with patients to receive an intravitreal injection of Aflibercept at the time of treatment.

ELIGIBILITY:
Inclusion Criteria

A subject must meet the following criteria to be eligible for inclusion in the study:

1. Signed Informed Consent.
2. Men and women ≥ 50 years of age.
3. Active primary subfoveal choroidal neovascularization (CNV) lesions secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by historical optical coherence tomographies (OCTs) and angiograms in the study eye.
4. CNV must be at least 50% of total lesion size by either previous or current angiogram.
5. ETDRS best-corrected visual acuity of: 20/25 to 20/320 (letter score of 73 to 25) in the study eye.
6. Willing, committed, and able to return for all clinic visits and complete all study related procedures.
7. At least one injection of Ranibizumab or Bevacizumab within 3 months of enrollment for active exudative AMD.
8. Active need for anti- vascular endothelial growth factor (anti-VEGF) therapy at study entry based on the following criteria:

   1. Presence of fluid by either optical coherence tomography (OCT) or clinical examination (further defined as intraretinal, cystoid, subretinal, worsening pigment epithelial detachment)
   2. Presence of new hemorrhage on clinical examination

Exclusion Criteria

A subject who meets any of the following criteria will be excluded from the study:

1. Any prior or concomitant therapy with another investigational agent to treat neovascular AMD in the study eye, except dietary supplements or vitamins.
2. Prior systemic anti-VEGF therapy, investigational or FDA/Health Canada approved, is only allowed up to 3 months prior to first dose, and will not be allowed during the study.
3. Presence of retinal pigment epithelial tears or rips involving the macula in the study
4. History of any vitreous hemorrhage within 4 weeks prior to Visit 1 in the study eye.
5. Presence of other causes of CNV, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, or multifocal choroiditis in the study eye.
6. History or clinical evidence of diabetic retinopathy, diabetic macular edema or any other vascular disease affecting the retina, other than AMD, in either eye.
7. Prior vitrectomy in the study eye.
8. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
9. Any history of macular hole of stage 2 and above in the study eye.
10. Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as it's unlikely to interfere with the injection.
11. Prior trabeculectomy or other filtration surgery in the study eye.
12. Uncontrolled glaucoma at baseline evaluation (defined as intraocular pressure ≥25 mmHg despite treatment with anti-glaucoma medication) in the study eye.
13. Active intraocular inflammation in either eye.
14. Active ocular or periocular infection in either eye.
15. Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
16. Any history of uveitis in either eye.
17. Active scleritis or episcleritis in either eye.
18. Presence or history of scleromalacia in either eye.
19. Aphakia or pseudophakia with absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet (YAG) posterior capsulotomy) in the study eye.
20. Previous therapeutic radiation in the region of the study eye.
21. History of corneal transplant or corneal dystrophy in the study eye.
22. Significant media opacities, including cataract, in the study eye which might interfere with visual acuity, assessment of safety, or fundus photography.
23. Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 52 week study period.
24. Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
25. Participation as a subject in any clinical study within the 12 weeks prior to Day 1.
26. Any systemic with an investigational agent in the past 3 months prior to Day 1.
27. The use of long acting intraocular steroids or photodynamic therapy in the 6 months prior to day 1.
28. Any history of allergy to povidone iodine.
29. Pregnant or breast-feeding women
30. Women of childbearing potential* who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

    * *Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rishi P Singh, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh RP, Srivastava SK, Ehlers JP, Silva FQ, Bedi R, Schachat AP, Kaiser PK. A single-arm, investigator-initiated study of the efficacy, safety, and tolerability of intravitreal aflibercept injection in subjects with exudative age-related macular degeneration previously treated with ranibizumab or bevacizumab (ASSESS study): 12-month analysis. Clin Ophthalmol. 2015 Sep 22;9:1759-66. doi: 10.2147/OPTH.S87043. eCollection 2015. PMID 26445522
- [Result] Singh RP, Srivastava S, Ehlers JP, Bedi R, Schachat AP, Kaiser PK. A single-arm, investigator-initiated study of the efficacy, safety and tolerability of intravitreal aflibercept injection in subjects with exudative age-related macular degeneration, previously treated with ranibizumab or bevacizumab: 6-month interim analysis. Br J Ophthalmol. 2014 Jun;98 Suppl 1(Suppl 1):i22-27. doi: 10.1136/bjophthalmol-2013-304798. PMID 24836866

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group: Subjects were included in the study if they met the following criteria: (1) active subfoveal choroidal neovascularization secondary to exudative Age-related Macular Degeneration (AMD) confirmed by fluorescein angiography (2) E-ETDRS vision of 25 to 80 letters (Snellen equivalent of ~20/25 to 20/320) (3) at least one prior injection of 1.25 mg bevacizumab or 0.5 mg ranibizumab (Avastin and Lucentis, respectively; Genentech Inc, South San Francisco, California, USA) within 3 months of enrollment, and (4) had an initial response on optical coherence tomography (OCT) defined as a decrease of retinal edema and/or subretinal fluid to anti-Vascular Endothelial Growth Factor (anti-VEGF) injections followed by recurrent increase in fluid on OCT (further defined as intraretinal, cystoid, subretinal fluid, or worsening pigment epithelial detachment) or the presence of a new hemorrhage on clinical examination.
Period: Overall Study
Arm/Group | Single Group
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 26 eyes, 01 eye per subject
Groups:
- Single Group: Subjects were included in the study if they met the following criteria: (1) active subfoveal choroidal neovascularization secondary to exudative AMD confirmed by fluorescein angiography (2) E-ETDRS vision of 25 to 80 letters (Snellen equivalent of ~20/25 to 20/320) (3) at least one prior injection of 1.25 mg bevacizumab or 0.5 mg ranibizumab (Avastin and Lucentis, respectively; Genentech Inc, South San Francisco, CA, USA) within 3 months of enrollment, and (4) had an initial response on optical coherence tomography (OCT) defined as a decrease of retinal edema and/or subretinal fluid to anti-VEGF injections followed by recurrent increase in fluid on OCT (further defined as intraretinal, cystoid, subretinal fluid, or worsening pigment epithelial detachment) or the presence of a new hemorrhage on clinical examination.
Arm/Group | Single Group
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 26
Region of Enrollment [Number; unit: participants]
  United States | 26
Length of time since diagnosis of exudative AMD [Mean (Standard Deviation); unit: months] | 14 (11)
Time since last injection prior to study enrollment [Mean (Standard Deviation); unit: days] | 50 (24)
Previous treatment [Count of Participants; unit: Participants]
  Previous treatment- Bevacizumab | 7
  Previous treatment- Ranibizumab | 17
  Previous treatment- Bevacizumab and Ranibizumab | 2
Average number of treatments prior to study entry [Mean (Standard Deviation); unit: injections] | 9.62 (6.58)
Average number of injections during study [Mean (Standard Deviation); unit: injections] | 7.92 (0.27)
E-ETDRS best-corrected visual acuity (BCVA) letter score [Mean (Standard Deviation); unit: E-ETDRS letters] — The scale provided is the Eletronic-Early Treatment in Diabetic Retinopathy Scale (E-ETDRS) best corrected visual acuity scale. This is a very common ophthalmology measurement tool and it is quite clear from its name. Values that are higher are considered better and values that are lower are considered worse. Minimum E-ETDRS was 24 E-ETDRS letters and maximum E-ETDRS was 80 E-ETDRS letters.
  E-ETDRS letters | 56.42 (17.04)
Best Corrected Visual Acuity Snellen equivalent [Mean (Full Range); unit: E-ETDRS letters] — The Snellen Equivalent is a numerical values from 90-0 with the higher value indicated better visual acuity
  E-ETDRS letters | 0.25 [0.06 to 0.8]
Central subfield thickness [Mean (Standard Deviation); unit: µm] | 304.08 (75.44)

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Subfield Thickness From Baseline at 12 Months
Description: The mean absolute change from baseline central subfield thickness at 12 months as measured by SDOCT
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Single Group
Number analyzed (Participants) | 26
µm | -50.3 (63.9)
Statistical Analysis 1: Comparison: Single Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Best-corrected Visual Acuity From Baseline at 12 Months
Description: The mean absolute change from baseline in best-corrected visual acuity score at 12 months as measured by Eletronic-Early Treatment in Diabetic Retinopathy Scale (E-ETDRS) protocol. There were no sub scales used. These are common methods for ophthalmology studies to report their findings. The scale provided is the Electronic-Early Treatment in Diabetic Retinopathy Scale (E-ETDRS) best corrected visual acuity scale. Values that are higher are considered better and values that are lower are considered worse. Minimum E-ETDRS was 24 E-ETDRS letters and maximum E-ETDRS was 80 E-ETDRS letters.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: E-ETDRS letters
Arm/Group | Single Group
Number analyzed (Participants) | 26
E-ETDRS letters | 9.2 (9.5)
Statistical Analysis 1: Comparison: Single Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change in Macular Volume From Baseline at 12 Months.
Description: Mean absolute change from baseline in macular volume at 12 months.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Single Group
Number analyzed (Participants) | 26
mm3 | -0.4 (1.0)
Statistical Analysis 1: Comparison: Single Group; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

4. Secondary Outcome: Change in Cube Average Thickness From Baseline at 12 Months
Description: Mean absolute change in cube average thickness as measured by SDOCT from baseline at 12 months.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Single Group
Number analyzed (Participants) | 26
µm | -11.9 (27.6)
Statistical Analysis 1: Comparison: Single Group; Test type: Superiority or Other; p = 0.038, t-test, 2 sided

5. Secondary Outcome: Percentage of Patients Who Gained Greater Than 15 Letters of Vision From Baseline at 12 Months.
Description: The percentage of patients who gained greater than 15 letters of vision from baseline to 12 months.
Time Frame: baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group
Number analyzed (Participants) | 26
Participants | 7

6. Secondary Outcome: Percentage of Patients Who Lost Greater Than 15 Letters of Vision From Baseline at 12 Months
Description: The percentage of patients who lost greater than 15 letters of vision from baseline at 12 months.
Time Frame: baseline and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group
Number analyzed (Participants) | 26
Participants | 0

7. Secondary Outcome: Percentage of Subjects Who Were 20/40 or Better at Month 12.
Description: Percentage of subjects who had vision acuity of 20/40 or better at month 12.
Time Frame: month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group
Number analyzed (Participants) | 26
Participants | 13

8. Secondary Outcome: Percentage of Subjects Who Were 20/200 or Worse at Month 12.
Description: Percentage of subjects who had visual acuity of 20/200 or worse at month 12.
Time Frame: month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group
Number analyzed (Participants) | 26
Participants | 3

ADVERSE EVENTS:
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Group (N=26)
Cataract progression (Eye disorders) | 1 — Patient began noticing a myopic shift, and the vision loss due to cataract progression was identified. The patient underwent uncomplicated phacoemulsification and lens implant placement with significant improvement in visual acuity.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Group (N=26)
Cataract progression (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
The drawbacks of this study included the small sample size and only 12 months of follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No